CLINICAL TRIAL: NCT02744534
Title: Targeted Fusion Biopsy of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Baowei Fei, PhD, EngD, Associate Professor and Georgia Cancer Coalition Distinguished Scholar, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00080287; R21CA176684 (NIH); R01CA156775 (NIH); R01CA204254 (NIH)
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Imaging Technology; Oncology; Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abnormalities found with FACBC PET-CT (Experimental): All participants with suspected recurrence of prostate cancer will have the FACBC PET-CT scan performed. Participants with abnormal FACBC PET-CT scan results will have a PET/ultrasound fusion targeted prostate biopsy followed a standard of care prostate biopsy.
  Interventions: Drug: FACBC PET-CT Scan; Procedure: Three-dimensional ultrasound-guided biopsy; Procedure: Standard transrectal ultrasound (TRUS) guided biopsy
- No abnormalities found with FACBC PET-CT (Active Comparator): All participants with suspected recurrence of prostate cancer will have the FACBC PET-CT scan performed. Participants without abnormal FACBC PET-CT scan results will have a standard of care prostate biopsy.
  Interventions: Drug: FACBC PET-CT Scan; Procedure: Standard transrectal ultrasound (TRUS) guided biopsy

INTERVENTIONS:
Drug: FACBC PET-CT Scan — One hour prior to scanning, participants will drink one glass (450 ml) of oral contrast to allow for better pictures of abdomen and pelvic organs. The participants will have their temperature taken before and after the injection of the FACBC. Blood pressure and pulse will be taken every 15 minutes during the PET scan.
  Participants will lie on a scanning bed and the bed will move slowly through the PET/CT scanner. This portion usually takes about one minute. Following this the FACBC will by administered by an intravenous (IV) catheter and the PET scan portion of the exam will begin. The table moves slowly through the scanner and many sets of PET-CT images are produced. When the imaging is complete, the scanner will send the results to a computer. The computer then generates a number of images that will be reviewed by a specially trained radiologist.
Procedure: Three-dimensional ultrasound-guided biopsy — A lubricated rectal probe will be inserted and a local anesthetic to numb the prostate will be administered. The ultrasound probe allows visualization of the prostate in two-dimensional (2D) images. The probe connects to a computer that will link to the FACBC PET-CT scan results that the participant has already had performed. These combined images will provide a three-dimensional (3D) image from the FACBC PET-CT scan previously obtained as well as real-time, 2D ultrasound images, resulting in an improved visualization tool to target the biopsy needle to a suspicious lesion.
  The needle tip position for each biopsy sample will be recorded on the real-time ultrasound images; this information allows the physician to either re-biopsy the same area for a follow-up examination or not to re-biopsy the same region if the original biopsy was negative.
  This biopsy process is estimated to take about 10 minutes.
  Other Names: Targeted prostate biopsy
  Arms: Abnormalities found with FACBC PET-CT
Procedure: Standard transrectal ultrasound (TRUS) guided biopsy — A lubricated ultrasound probe of about 2.5 cm in diameter is gently inserted into the rectum and a local anesthetic to numb the prostate is administered. The ultrasound probe allows visualization of the prostate in two-dimensional (2D) images and allows for the placement of a biopsy needle that collects samples of the prostate. Usually, a total of 12 biopsy specimens are collected. The procedure takes about 20 minutes. This TRUS-guided biopsy is considered as the standard method for prostate cancer diagnosis.
  Other Names: Standard prostate biopsy

SUMMARY:
The purpose of this study is to see if using Positron Emission Tomography (PET) scan and transrectal ultrasound (TRUS) guided biopsy together (creating a 3-dimensional ultrasound) will detect prostate cancer more accurately than the standard 2-dimensional approach which uses only the TRUS to guide the biopsy.

DETAILED DESCRIPTION:
The objective of the proposed study is to evaluate a molecular image directed, three-dimensional (3D) ultrasound guided biopsy system in human patients. Prior studies have shown that Positron Emission Tomography (PET)/Computed Tomography (CT) imaging with the PET molecular imaging agent, a synthetic amino acid, anti-1-amino-3-[18F]fluorocyclobutane-1- carboxylic acid (FACBC), is more sensitive than the FDA-approved prostate specific membrane antigen single-photon emission computed tomography (SPECT) radiotracer in prostate cancer detection. FACBC images showed higher focal uptake in tumor foci than in normal prostate and thus could be ideal information to direct targeted biopsy of the prostate. This targeted biopsy system has a unique feature that PET/CT images can be registered with 3D ultrasound images, as a result, a suspicious PET lesion is superimposed over the real-time ultrasound data; and the fused image is then used to direct biopsy needles to tumor targets.

The hypothesis of the study is that PET/ultrasound fusion targeted biopsy can detect more cancer per core than the standard 12-core TRUS guided biopsy.

The specific aims include:

1. To perform PET/CT directed, 3D ultrasound-guided biopsy and determine if fusion targeted biopsy can detect more cancers than 2D transrectal ultrasound (TRUS)-guided biopsy
2. To develop the workflow for performing deformable registration and fusion of PET/CT and 3D ultrasound images of human patients

Thirty six patients, who have suspicion of recurrent prostate cancer after definitive therapy such as radiotherapy, will be recruited into this study. At least half of the patients will have positive imaging findings and will undergo 2D TRUS-guided biopsy as well as PET/ultrasound fusion biopsy. The proposed study will be the first-in-human trial that uses PET/CT imaging to direct 3D ultrasound-guided biopsy of the prostate. The multimodality imaging approach will combine the high sensitivity from PET and real-time information from ultrasound for improved cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Have been originally diagnosed with prostate carcinoma and have undergone definitive non-prostatectomy therapy for localized disease
* There is suspicion of recurrent prostate carcinoma as defined by: Older American Society for Radiation Oncology (ASTRO) criteria of three consecutive rises of prostate-specific antigen (PSA) or earlier if clinically appropriate, and/or nadir + 2.0 ng/ml (Radiation Therapy Oncology Group (RTOG)-ASTRO Phoenix criteria)
* Able to provide written informed consent

Exclusion Criteria:

* Cryotherapy, external beam radiation, or high intensity focused ultrasound (HIFU) within the past year
* Brachytherapy within the past two years (to rule out a transient rise in PSA)
* Prostate biopsy within the past month (to decrease a false positive result due to inflammation)
* Not otherwise eligible for prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baowei Fei, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital and the Winship Cancer Institute in Atlanta, Georgia from November 2015 to April 2017. All study procedures were completed by March 31, 2018.
Pre-assignment Details: Participants with abnormal anti-1-amino-3-[18F]fluorocyclobutane-1- carboxylic acid (FACBC) positron emission tomography (PET)-CT scans were to have both targeted and template biopsies while those with normal FACBC PET-CT scans would have only the standard of care template biopsy. None of the study participants had a normal FACBC PET-CT scan.
Groups:
- Targeted Biopsy and Template Biopsy: Study participants with abnormal FACBC PET-CT scans received a fluciclovine PET ultrasound fusion targeted biopsy and a template (standard of care) biopsy to test for recurrent prostate cancer.
Period: Overall Study
Arm/Group | Targeted Biopsy and Template Biopsy
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Targeted Biopsy and Template Biopsy: Study participants with abnormal FACBC PET-CT scans received a targeted biopsy and a template (standard of care) biopsy to test for recurrent prostate cancer.
Arm/Group | Targeted Biopsy and Template Biopsy
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
Prostate-Specific Antigen (PSA) prior to PET scan [Mean (Standard Deviation); unit: ng/ml] | 7.4 (6.8)
Initial therapy [Count of Participants; unit: Participants]
  Radiotherapy | 9
  Non-radiotherapy (cryotherapy) | 3
  Mixed therapy | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cores Positive for Cancer
Description: The cancer detection rate per core was compared between the targeted prostate biopsy and standard of care prostate biopsy.
Time Frame: Two weeks
Population: All 21 participants are included in the analysis, and all participants had both types of biopsies performed. The total number of core samples taken during biopsy are given as the overall number of participants analyzed and the percentage of these core samples that tested positive for prostate cancer are given as the outcome measure data.
Measure: Number; unit: percentage of positive core samples
Units Other Than Participants: Prostate biopsy core samples
Groups:
- Targeted Biopsy: Fluciclovine defined targets were biopsied using the 3-D visualization and navigation platform to guide the biopsy needle and record its path.
- Standard Biopsy: The standard transrectal ultrasound guided biopsy collects 2 cores per region (when possible) from 6 standard regions of the prostate.
Arm/Group | Targeted Biopsy | Standard Biopsy
Number analyzed (Participants) | 21 | 21
Number analyzed (Prostate biopsy core samples) | 125 | 246
percentage of positive core samples | 32.0 | 4.5

ADVERSE EVENTS:
Time Frame: The time period for collecting adverse events was from the the time of the FACBC PET-CT scan until 7 days after the scan. Since 95% of the ligand used during the scan is eliminated within 7 days, any events beyond 7 days after the scan were not considered to be adverse events due to study procedures.
Description: This study only collected adverse events that were a significant shift from baseline and which could be attributed to the radiotracer injection and not the patient's prior medical condition. No adverse events due to the study procedures were anticipated.
Groups:
- Targeted Biopsy; Template Biopsy: Study participants with abnormal FACBC PET-CT scans received a targeted biopsy and a template (standard of care) biopsy to test for recurrent prostate cancer.
Arm/Group | Targeted Biopsy | Template Biopsy
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02744534/Prot_SAP_000.pdf